CLINICAL TRIAL: NCT01807481
Title: A Prospective,Single-arm,Multicenter Study to Evaluate the Efficacy and Safety of Mircera in Peritoneal Patients Who Already Had Been Treated With ESA
Brief Title: Phase IV Study to Evaluate the Efficacy and Safety of Mircera in PD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim Dae Joong, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2011-10-131
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: PD
Keywords: Mircera; PD; Maitenance
MeSH Terms: interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mircera Arm (Experimental): Once Monthly Mircera
  Interventions: Drug: Mircera

INTERVENTIONS:
Drug: Mircera — Once Monthly Mircera

SUMMARY:
The primary objective of study is to evaluate the no of patients which maintain the Hb level between 9.0 ~ 12.0 g/dl during the evaluation period

DETAILED DESCRIPTION:
The secondary objective of study is

* No of patients with mean Hb level of +/-1.0g/dl difference from the baseline Hb
* Incidence of RBC transfusion during the titration and evaluation periods
* Mean Hb during the total study period
* Intrapatient Hb variability (mean within-patient standard deviation for Hb)
* Frequency of Micera dose level
* safety

ELIGIBILITY:
Inclusion criteria:

* 1.≥18 yr of age
* 2.peritoneal dialysis for ≥12wk before screening and during baseline period
* 3.weekly Kt/V ≥1.8 for PD patients
* 4.Baseline Hb concentration between 9.0 and 12.0g/dl(mean of the monthly Hb values determined in month -2 and -1)
* 5.stable baseline Hb concentration(defined as an absolute difference ≤2g/dl between the Hb values determined in month -2 and -1)
* 6.continuous subcutaneous maintenance epoetin or darbepoetin therapy for at least 2 months before screening and during baseline period
* 7.adequate iron status defined as serum ferritin ≥ 100ng/ml or transferrin saturation≥20%(mean of two values deteremined in month -2 and -1)

Exclusion criteria:

* 1.Overt gastrointestinal bleeding or any other bleeding episode necessitating transfusion wihin 2 months before screening during baseline pereiod
* 2.RBC transfusions within 2 months before screening or during baseline period
* 3.nonrenal causes of anemia(e.g folic acid or vitamin B12 deficiency,hemolysis)
* 4.acute infection or chronic, uncontrolled or symptomatic inflammatory disease(e.g rhematoid arthritis,systemic lupus erythematosus)
* 5.C-reactive protein>30mg/dl
* 6.poorly controlled hypertension necessitating interruption of epotien or darbepoetin in the 6 months before screening
* 7.platelets > 500X109/L
* 8.pure red cell aplasia
* 9.chronic congestive heart failure(New Yorj Heart Association class IV)
* 10.Myocardial infarction,severe or unstable coronary artery disease,stroke,severe liver disease within the 3months before screening or during baseline
* 11.Life expectancy < 12months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hemoglobin 10~12 g/dl | Visit 0 ~ visit 10 (10 months)
  The primary objective of this study is to evaluate the no of patients which maintain the Hb-level between 10.0~13.0 g/dL during the evaluation period

SECONDARY OUTCOMES:
Hemoglobin stability, Dose adjustment | Visit0~Visit 10 (10 Months)
  Incidence of RBC transfusion during the titration and evaluation periods Mean Hb during the total study period Intrapatient Hb variability (mean within patient standard deviations for Hb) Comparison between baseline and evaluation period mean Hb level Frequency of dose adjustments Safety

CONTACTS AND LOCATIONS:
Overall Officials: Dae Joong Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea